CLINICAL TRIAL: NCT00333580
Title: Veteran-Centered Outcomes Using Qualitative and Quantitative Methods
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: O4052-X; IRB 03-2006 (Other: University of Florida IRB)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Spinal Cord Injury; Stroke
Keywords: Ethnography; Psychometrics; Qualitative Research
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The purpose of this study is to modify and develop measures that reflect outcomes that are relevant to recovering Veterans and are sensitive to improvements resulting from innovative gait interventions.

DETAILED DESCRIPTION:
Existing clinically-generated measures, in general, have been developed independent of input from Veterans. The purpose of this collaborative study is to take advantage of qualitative and quantitative expertise from the Gainesville, Florida, Rehabilitation Outcomes Research Center (RORC) with state-of-the-art gait intervention research being conducted at the Gainesville, Brain Rehabilitation Research Center (BRRC) and Cleveland, Functional Electrical Stimulation Center (FESC). Three interventions have received considerable attention for their demonstrated promise in improving gait and mobility in individuals with spinal cord injury and stroke; 1) manually assisted locomotor training (MLT), 2) robotic assisted locomotor training (RLT)and 3) functional electrical stimulation assisted gait training (FES-GT). These interventions will be the basis for improving existing outcome measures and developing new outcome measures. The process of developing and evaluating valid outcome measures requires four phases of development. This study encompasses Phases I and II. Phase I (Year 1 of grant)will involve completing qualitative research studies to identify constructs reflecting the impact of MLT, RLT and FES-GT on Veterans. Data will be systematically collected using ethnographic field observations and in depth, semi-structured interviews. Phase II (Year 2) will involve using the identified constructs to develop item banks for Veterans-centered outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stroke and patients with incomplete spinal cord injuries currently enrolled in locomotor/gait training studies at the VA BRain Rehabilitation Research Center, Gainesville, FL and the VA Functional Electrical Stimulation Center, Cleveland, Ohio, Competence for inclusion in the treatment intervention study (and the present study) is passing the 3-step command component of the Mini Mental Status Exam.

Exclusion Criteria:

* Unable to pass the 3-step command component of the Mini-Mental Exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veteran and non-veteran male/females with stroke or incomplete spinal cord injury currently enrolled in locomotor/gait training studies.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Narrative from qualitative interviews and ethnographic analysis of video diaries. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

REFERENCES:
- [Result] Hannold EM, Hanjian JM, Jordan MM, Roach MJ, Velozo CA. Using veterans' perspectives to enhance rehabilitation outcome measures: value of qualitative methods. J Rehabil Res Dev. 2008;45(1):xi-xv. No abstract available. PMID 18566921
- [Result] Jordan MM, Berkowitz D, Hannold E, Velozo CA, Behrman AL. Thinking through every step: how people with spinal cord injuries relearn to walk. Qual Health Res. 2013 Aug;23(8):1027-41. doi: 10.1177/1049732313494119. Epub 2013 Jun 17. PMID 23774628